CLINICAL TRIAL: NCT06904950
Title: Pilot Trial of Nightmare Deconstruction and Reprocessing, a Novel Treatment for PTSD-Related Nightmares and Insomnia
Brief Title: Nightmare Deconstruction and Reprocessing Pilot
Acronym: NDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patricia Spangler, Research Assistant Professor, Uniformed Services University of the Health Sciences
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSY-88-9157
Record Dates: First submitted 2021-09-28; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Nightmare
Keywords: Nightmares; Sleep disturbance; Posttraumatic
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: Single-arm pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nightmare Deconstruction and Reprocessing (NDR) (Experimental): Eight-session exposure-based treatment for posttraumatic nightmares and insomnia.
  Interventions: Behavioral: Nightmare Deconstruction and Reprocessing

INTERVENTIONS:
Behavioral: Nightmare Deconstruction and Reprocessing — Eight-sessions that include 1 session of psychoeducation and treatment orientation and 7 sessions of NDR. NDR consists of three stages: (1) nightmare image deconstruction, (2) meaning making and reprocessing of cognition and emotions related to images, (3) rescripting new dream images and rehearsal of new images.

SUMMARY:
This is a single-arm, multisite (2 sites) pilot trial that is evaluating Nightmare Deconstruction and Reprocessing (NDR) for treating posttraumatic nightmares and insomnia in up to 30 military service members and veterans. Study aims are to test NDR's plausibility and tolerability and to test methodologic feasibility of collecting heart rate variability (HRV), electrodermal activity (EDA), and actigraphy data via a wristband device and peripheral blood samples within a pre-specified circadian window. Treatment consists of 8 sessions over 8 weeks. Participants are assessed at study visits 0, 1, and 7 and 1-month follow-up. Psychometric assessments include the Disturbing Dreams and Nightmare Severity Index, Pittsburgh Sleep Quality Index, and Clinician-Administered PTSD Scale for DSM-5.

DETAILED DESCRIPTION:
The current study is testing NDR, a three-stage treatment that integrates exposure, reprocessing, and rescripting of nightmare images to alleviate nightmare and insomnia severity. Study aims are to test NDR's plausibility and tolerability and to test the methodologic feasibility of collecting daily HRV, EDA, and actigraphy data via the E4 wristband as well as peripheral blood samples for assay at three time points. Participants are active duty military or veterans (N = 30) ages 18 to 64 with posttraumatic nightmares and insomnia. Participants undergo 8 NDR treatment visits over 8 weeks and complete a 1-month follow-up. Psychometric measures of nightmare (Disturbing Dreams and Nightmare Severity Index) and insomnia (Pittsburgh Sleep Quality Index) are administered at each visit. Objective measurement of sleep disturbance is done via the Empatica E4 wristband. In-session distress is measured using the 1-item Subjective Units of Distress Scale (SUDS), and E4 HRV and EDA data during exposure to nightmare images. BDNF, IL-2, IL-6, and TNF alpha are being assayed from blood samples taken immediately after Visit 0 (baseline), Visit 1 (first in-session exposure to nightmare images), and Visit 7 (final in-session exposure to nightmares). To control for circadian factors regulating the expression of BDNF and inflammatory cytokines, all blood samples are collected between 0900 and 1200.

ELIGIBILITY:
Inclusion Criteria:

* Active duty servicemembers and DEERS-eligible veterans
* DDNSI score ≥ 10
* PSQI score > 5

Exclusion Criteria:

* Current imminent risk of suicide
* Psychotic or bipolar disorders
* Untreated moderate to severe sleep apnea/hypopnea, circadian rhythm disorders, or narcolepsy
* Current use of prazosin for nightmares
* Self-reported alcohol use > 4x/ week and > 3 drinks per occasion
* Concurrent evidence-based or experimental treatment directly targeting nightmares, insomnia, or PTSD
* Initiation of or change in psychotropic medications for PTSD, nightmares, insomnia, depression, or anxiety in the past 8 weeks
* Inability to recall nightmare content
* Inability to comply with requirement to wear E4 wristband and upload daily

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Disturbing Dream and Nightmare Severity Index (DDNSI) | Up to16 weeks, starting with screening, then weekly through the treatment period (8 weeks), and at follow-up (1 month)
  5-item instrument used to assess nightmare severity and distress, scored by adding nights/per week (0 to 7) + nightmares/week +Q3 (0 to 4 scale) +Q4 (0 to 6 scale) + Q5 (0 to 6 scale). Higher scores indicate greater symptom severity. >10 indicates nightmare disorder and was used as the inclusion cutoff for the study.
Pittsburgh Sleep Quality Index (PSQI) | Up to16 weeks, starting with screening, then weekly through the treatment period (8 weeks), and at follow-up (1 month)
  19-item instrument with 7 components that are scored on a 0-3 Likert-type scale, with higher scores indicating poorer sleep quality. >5 indicates significant sleep disturbance and was used an inclusion cutoff for the study.

SECONDARY OUTCOMES:
Clinician-Administered PSTD Scale for DSM-5 (CAPS-5) | Up to16 weeks, starting with screening, then at the end of the treatment period (8 weeks), and at follow-up (1 month).
  30-item structured clinical interview assessing DSM-5 diagnostic criteria for PTSD. Symptoms assessed on a 5-point scale (0-4), with higher scores indicating greater symptom severity.

OTHER OUTCOMES:
In-Session Heart Rate (HR) | Approximately 10 weeks, data collected continuously (23 hours per day) during the treatment period (8 weeks) and 2 weeks into the follow-up period.
  HR was collected with the E4 wristband to assess pre- to post-treatment change in response to in-session exposure to nightmare images.
In-session Electrodermal Activity (EDA) | Approximately 10 weeks, data collected continuously (23 hours per day) during the treatment period (8 weeks) and 2 weeks into the follow-up period.
  EDA was collected with the E4 wristband to assess pre- to post-treatment change in response to in-session exposure to nightmare images.
Brain-derived neurotropic factor (BDNF) | 8 weeks: blood samples taken immediately after Visit 0 and Visit 1 (week 1) and immediately after Visit 7 (week 8)
  BDNF was assayed from blood samples to evaluate pre- to post-treatment change in expression in response to exposure to nightmare images.
Inflammatory cytokines | 8 weeks: blood samples taken immediately after Visit 0 and Visit 1 (week 1) and immediately after Visit 7 (week 8)
  Inflammatory cytokines were assayed from blood samples to evaluate pre- to post-treatment change in expression in response to exposure to nightmare images. All blood samples taken between 0900 and 1200 to control for circadian variability in expression.
Sleep Actigraphy Data | Approximately 10 weeks, data collected continuously (23 hours per day) during the treatment period (8 weeks) and 2 weeks into the follow-up period.
  Actigraphy data was collected with the E4 wristband to assess change in sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia T Spangler, PhD, Principal Investigator — Uniformed Services University and Henry M Jackson Foundation
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description of study — https://www.cstsonline.org/research/active-research-studies
- See also: Study recruitment survey — https://redcap.hjf.org/surveys/?s=YEYHM97M4C
- See also: Study Facebook page — https://www.facebook.com/NDRforPTSD